CLINICAL TRIAL: NCT00969982
Title: Mifepristone and Misoprostol Versus Misoprostol Alone for Mid-trimester Termination of Pregnancy (14 - 21 Weeks LMP): A Randomized-controlled Double-blinded Trial
Brief Title: Mifepristone Plus Misoprostol Versus Misoprostol Alone for 2nd Trimester Abortion (14 - 21 Weeks Last Menstrual Period (LMP))
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.4.1
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Abortion, Induced
Keywords: Pregnancy termination; abortion; medical abortion; 2nd trimester; mifepristone; misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mifepristone+misoprostol (Experimental): 200 mg mifepristone followed by 800 mcg buccal misoprostol repeated every 3 hours until complete abortion or maximum of 10 doses within 48 hours (maximum 5 doses per 24 hours).
  Interventions: Drug: mifepristone+misoprostol
- misoprostol (Active Comparator): Placebo resembling mifepristone followed 24 hours later by 800 mcg buccal misoprostol repeated every 3 hours until complete abortion up to a maximum of 10 doses within 48 hours (maximum 5 doses per 24 hours).
  Interventions: Drug: misoprostol+placebo

INTERVENTIONS:
Drug: mifepristone+misoprostol — single dose of 200 mg mifepristone followed 24 hours later by 800 mcg misoprostol administered buccally and repeated every 3 hours for a maximum of 5 doses per 24 hours up to 48 hours.
  Arms: mifepristone+misoprostol
Drug: misoprostol+placebo — placebo resembling mifepristone followed 24 hours later by 800 mcg buccal misoprostol repeated every 3 hours for a maximum of 5 doses per 24 hours up to 48 hours.
  Arms: misoprostol

SUMMARY:
The primary goal of this study is to determine the clinical advantage of pre-treatment with mifepristone in second trimester misoprostol induction abortion. This will be a randomized controlled double-blinded trial of 120 women in each country comparing misoprostol alone to mifepristone plus misoprostol for second trimester (14-21 weeks' LMP) medical abortion.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 21 weeks gestation, based on menstrual history and clinical exam (with or without ultrasound)
* Meet legal criteria to obtain abortion
* Present with closed cervical os and no vaginal bleeding
* Live fetus at time of presentation for service
* Have no contraindications to study procedures, according to provider
* Be able to consent to procedure, either by reading consent document or by having consent document read to her
* Be willing to follow study procedures

Exclusion Criteria:

* Known previous transmural uterine incision
* Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
* Any contraindications to vaginal delivery, including placenta previa
* Presentation in active labor (defined as moderate to severe contractions every 10 minutes or less)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Rate of successful abortion: defined as complete evacuation using study drug without recourse to any additional intervention. | 48 hours
Induction-to-abortion interval: defined as time elapsed between administration of the first misoprostol dose until expulsion of the fetus. | 48 hours

SECONDARY OUTCOMES:
Provision of additional interventions to manage excessive blood loss | from start of treatment until discharge
Any heavy bleeding, uterine rupture, or infection requiring additional treatment | start of treatment until discharge
Total dose of misoprostol. | Assessed at time of complete abortion with study drug alone or when total maximum dose given.
Pain experienced by the woman as self-reported. | Assessed during exit interview.
Women's acceptability of the assigned method | Assessed at exit interview

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, Principal Investigator — Gynuity Health Projects
Locations (2):
- Municipal Clinical Hospital, Chishinau, Moldova
- La Rabta Maternity Hospital, Tunis, Tunisia

REFERENCES:
- [Derived] Dabash R, Chelli H, Hajri S, Shochet T, Raghavan S, Winikoff B. A double-blind randomized controlled trial of mifepristone or placebo before buccal misoprostol for abortion at 14-21 weeks of pregnancy. Int J Gynaecol Obstet. 2015 Jul;130(1):40-4. doi: 10.1016/j.ijgo.2015.02.023. Epub 2015 Apr 11. PMID 25896965